CLINICAL TRIAL: NCT05197647
Title: Cohort Study for the Assessment of Long-term Impact of COVID-19 Among Mild COVID-19 Patients in Brazil
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Moinhos de Vento (Other)
Responsible Party: Sponsor
Other Study IDs: Pos-COVID Brasil 2
Record Dates: First submitted 2022-01-14; First posted 2022-01-19 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; Quality of Life; Disability Physical; Disabilities Mental
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with mild COVID-19: Patients with symptomatic COVID-19 disease not requiring hospitalization.
  Interventions: Other: Patients with symptomatic COVID-19 disease not requiring hospitalization.

INTERVENTIONS:
Other: Patients with symptomatic COVID-19 disease not requiring hospitalization. — Patients with symptomatic COVID-19 disease not requiring hospitalization.

SUMMARY:
The present prospective cohort study aims to assess factors associated with of one-year health-related quality of life and physical, cognitive and mental health outcomes among adult patients with mild COVID-19. Adult patients with symptomatic COVID-19 not requiring hospitalization will be followed through structured and centralized telephone interviews performed at 1, 3, 6, 9 and 12 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Positive polymerase chain reaction (PCR) test for SARS-CoV-2;
* At least one of the following symptoms: fever, cough, sneezing, dyspnea, fatigue, smell alteration, rhinorrhea, sore throat, myalgia, arthralgia, diarrhea;
* Outpatient COVID-19 care at the moment of enrollment (without indication for in-hospital care).

Exclusion Criteria:

* Severe comorbidity with life expectancy less than 3 months;
* Absence of proxy for patients with communication difficulties;
* Absence of telephone contact;
* Refusal or withdrawal of agreement to participate;
* Previous enrollment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients survivors with proven mild symptomatic COVID-19 disease not requiring hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 1085 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
One-year utility score of health related quality of life | The outcome will be assessed 12 months after enrollment.
  The outcome will be assessed using the Brazilian version of the Euroqol-5D-3L (EQ-5D3L) questionnaire. The utility score derived from the EQ5D-3L ranges from 0 (death) to 1 (perfect health).

SECONDARY OUTCOMES:
Utility score of health related quality of life at 3, 6, and 9 months | The outcome will be assessed at 3, 6, and 9 months after enrollment.
  The outcome will be assessed using the Brazilian version of the Euroqol-5D-3L (EQ-5D3L) questionnaire. The utility score derived from the EQ5D-3L ranges from 0 (death) to 1 (perfect health).
Incidence of all-cause mortality | The outcome will be assessed at 1, 3, 6, 9, and 12 months after enrollment.
  Incidence of all-cause mortality
Incidence of major cardiovascular events | The outcome will be assessed at 3, 6, 9, and 12 months after enrollment.
  Incidence of major cardiovascular events (composite endpoint of non-fatal stroke, non-fatal acute myocardial infarction, or cardiovascular death)
Incidence of hospitalizations | The outcome will be assessed at 1, 3, 6, 9, and 12 months after enrollment.
  Incidence of all-cause hospitalizations
Prevalence of prolonged COVID-19 symptoms | The outcome will be assessed at 1, 3, 6, 9, and 12 months after enrollment.
  Prevalence of prolonged COVID-19 symptoms defined as presence of dyspnea, cough, fatigue, muscular weakness, chest discomfort, joint pain, anosmia, hair loss, brain fog, insomnia, among others)
Prevalence of cognitive dysfunction | The outcome will be assessed at 3, 6, 9, and 12 months after enrollment.
  Prevalence of cognitive dysfunction as assessed by the Telephone Interview for Cognitive Status (TICS-m; scores ranging from 0 to 50 with lower scores indicating worse cognition).
Prevalence of anxiety and depression symptoms | The outcome will be assessed at 3, 6, 9, and 12 months after enrollment.
  Prevalence of anxiety and depression symptoms as assessed by the Hospital Anxiety and Depression Scale (anxiety and depression scores range from 0 to 21, with higher scores indicating worse symptoms).
Prevalence of posttraumatic stress disorder symptoms | The outcome will be assessed at 3, 6, 9, and 12 months after enrollment.
  Prevalence of posttraumatic stress disorder symptoms as assessed by the Impact Event Scale-6 (scores range from 0 to 24 with higher scores indicating worse symptoms).
Physical functional status | The outcome will be assessed at 3, 6, 9, and 12 months after enrollment.
  Physical functional status as assessed by the modified Barthel index (score ranges from 0 to 100; higher scores indicate less functional dependence).
Instrumental Activities of Daily Living | The outcome will be assessed at 3, 6, 9, and 12 months after enrollment.
  The outcome will be assessed using the Lawton & Brody Instrumental Activities of Daily Living Scale (the score ranges from 0 to 8, with higher scores indicating less dependence).
Incidence of return to work or study | The outcome will be assessed at 3, 6, 9, and 12 months after enrollment.
  Incidence of return to work or study among patients that were working or studying at the moment of COVID-19 diagnosis.
Incidence of new symptomatic COVID-19 infection | The outcome will be assessed at 3, 6, 9, and 12 months after enrollment.
  Incidence of new symptomatic COVID-19 infection defined as recurrence of COVID-19-related symptoms with a positive PCR test for SARS-CoV-2 90 days after the index infection.

CONTACTS AND LOCATIONS:
Overall Officials: Regis Rosa, MD, PhD, Principal Investigator — Hospital Moinhos de Vento
Locations (14):
- Brazil (14):
  - Clinica Silvestre Santé, Rio Branco, Acre
  - Hospital Enseada Prime, Vitória, Espírito Santo
  - Hospital do Coração do Mato Grosso do Sul, Campo Grande, Mato Grosso do Sul
  - Hospital Metropolitano Célio de Castro, Belo Horizonte, Minas Gerais
  - Instituto Horizonti, Belo Horizonte, Minas Gerais
  - Hospital Universitário de Ponta Grossa, Ponta Grossa, Paraná
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital Vila Nova, Porto Alegre, Rio Grande do Sul
  - Instituto Procardio, Joinville, Santa Catarina
  - Hospital Leo Orsi, Itapetininga, São Paulo
  - Hospital de Clínicas de Ribeirão Preto, Ribeirão Preto, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo, São Paulo
  - Hospital do Coração, São Paulo, São Paulo
  - Hospital Santa Paula, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided
The authors encourage interested parties to contact the corresponding author with data sharing requests, including for access to additional unpublished data.

REFERENCES:
- [Background] Rover MM, Trott G, Scolari FL, Silva MMDD, Souza D, Santos RDRMD, Dagnino APA, Mesquita Neto J, Estivalete GP, Kozesinski-Nakatani AC, Marcolino MS, Barreto BB, Schvartzman PR, Antonio ACP, Robinson CC, Falavigna M, Biolo A, Polanczyk CA, Rosa RG. Health-Related Quality of Life and Long-Term Outcomes after Mildly Symptomatic COVID-19: The Post-COVID Brazil Study 2 Protocol. Arq Bras Cardiol. 2023 Sep;120(9):e20220835. doi: 10.36660/abc.20220835. English, Portuguese. PMID 37851732